CLINICAL TRIAL: NCT03893552
Title: Upper Airway Stability During Wakefulness and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, ALBDEWI Mohamad Ammar, Phd studant, Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Study 2015/01OCT/521
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea Syndromes; Snoring
Keywords: Negative expiratory pressure, sleep apnea, Snoring, Sleep-disordered breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with sleep disordered breathing symptoms (Experimental): Patients referring to the clinic of sleep disorders will be asked to participate in this study. A negative expiratory pressure will be applied via a cough-assist attached to a facial mask.
  Interventions: Device: Negative expiratory pressure

INTERVENTIONS:
Device: Negative expiratory pressure — Using a cough assist, a negative expiratory pressure will be applied while recording the respiratory flow in patients suffering from sleeping disorders or snoring.

SUMMARY:
Negative expiratory pressure is a technique that has been the focus of many studies in the last few years.

Airway response to the application of a negative expiratory pressure (NEP) can be used to detect the presence of upper airway collapsibility. In normal subjects, an increase in expiratory flow is observed while in patients with collapsible upper airway, the flow will show a transient decrease due to airway collapse.

The objectives of this study will be initially to investigate the diagnostic utility of this technique as a noninvasive measurement of the stability of the upper airway in sleep-related breathing disorders. Secondly, we aim to see the sites of airway obstructions, discovered by NEP, through nasal endoscopy. Finally, we aim at testing the utility of NEP technique in the evaluation of therapeutic response. For this purpose, we will apply it in patients before and after airway stabilization interventions like ENT surgery, oropharyngeal exercises, orthodontic mandibular advancement electrical stimulation of the hypoglossal nerve.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Patients with COPD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Measure of Flow limitation during NEP application | measurement done immediately after inclusion, one time
  see above, using pneumotachograph